CLINICAL TRIAL: NCT06606314
Title: Specified Drug-use Surveillance of Fabhalta Capsules (Paroxysmal Nocturnal Hemoglobinuria, CLNP023C11401)
Brief Title: Specified Drug-use Surveillance of Fabhalta Capsules
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CLNP023C11401
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Paroxysmal Nocturnal Hemoglobinuria
Keywords: paroxysmal nocturnal hemoglobinuria; PNH; Fabhalta
MeSH Terms: conditions — Hemoglobinuria, Paroxysmal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
This is a multicenter, single-arm, non-interventional study (NIS) with a central registration system and an all-case surveillance system. The observation period is 48 weeks after the start of treatment with Fabhalta.

DETAILED DESCRIPTION:
The observation period will be 48 weeks after the start of treatment with Fabhalta.

For patients in whom treatment with Fabhalta is discontinued within 48 weeks after the start of the treatment, adverse events occurring by the last day of the treatment + 30 days and concomitant drugs will be monitored and recorded in CRFs.

ELIGIBILITY:
Inclusion Criteria:

All patients who received Fabhalta.

·

Exclusion Criteria:

Patients receiving Fabhalta for an unapproved indication under the Clinical Trials Act or GCP.

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients who received Fabhalta.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-18 (Actual); Primary Completion 2028-09-30 (Estimated); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Occurrence status of infections. | 48weeks
  Type, incidence, seriousness, severity, clinical course, factors affecting onset (status of vaccination, name of vaccine administered, complications, baseline white blood cell count/neutrophil count, etc.), and causative organism (including serotype) of adverse events/adverse drug reactions of infections during the treatment period.

SECONDARY OUTCOMES:
Occurrence status of serious hemolysis after discontinuation of Fabhalta. | 48weeks
  Number of patients with serious hemolysis after discontinuation of Fabhalta.
Occurrence status of adverse events and adverse drug reactions. | 48weeks
  Incidence of adverse events and adverse drug reactions during the treatment period.
Incidence of breakthrough hemolysis and change of hemolysis-related markers and status of red blood cell transfusion-free. | 48weeks
  Incidence of breakthrough hemolysis per year and change over time in hemolysis-related markers (LDH, Hb, etc.) and status of red blood cell transfusion-free up to Week 48.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (73):
- Japan (73):
  - Novartis Investigative Site, Handa, Aichi-ken
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Okazaki, Aichi-ken
  - Novartis Investigative Site, Toyohashi, Aichi-ken
  - Novartis Investigative Site, Toyota, Aichi-ken
  - Novartis Investigative Site, Hachinohe, Aomori
  - Novartis Investigative Site, Funabashi, Chiba
  - Novartis Investigative Site, Kashiwa, Chiba
  - Novartis Investigative Site, Matsuyama, Ehime
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Kurume, Fukuoka
  - Novartis Investigative Site, Aizu-Wakamatsu, Fukushima
  - Novartis Investigative Site, Kohriyama, Fukushima
  - Novartis Investigative Site, Maebashi, Gunma
  - Novartis Investigative Site, Fukuyama, Hiroshima
  - Novartis Investigative Site, Hakodate, Hokkaido
  - Novartis Investigative Site, Sapporo, Hokkaido
  - Novartis Investigative Site, Amagasaki, Hyōgo
  - Novartis Investigative Site, Ashiya, Hyōgo
  - Novartis Investigative Site, Himeji, Hyōgo
  - Novartis Investigative Site, Kobe, Hyōgo
  - Novartis Investigative Site, Nishinomiya, Hyōgo
  - Novartis Investigative Site, Tsukuba, Ibaraki
  - Novartis Investigative Site, Kanazawa, Ishikawa-ken
  - Novartis Investigative Site, Morioka, Iwate
  - Novartis Investigative Site, Sakaidechō, Kagawa-ken
  - Novartis Investigative Site, Kanoya, Kagoshima-ken
  - Novartis Investigative Site, Isehara, Kanagawa
  - Novartis Investigative Site, Yokohama, Kanagawa
  - Novartis Investigative Site, Kyoto, Kyoto
  - Novartis Investigative Site, Uji, Kyoto
  - Novartis Investigative Site, Ōsaki, Miyagi
  - Novartis Investigative Site, Miyazaki, Miyazaki
  - Novartis Investigative Site, Nobeoka, Miyazaki
  - Novartis Investigative Site, Matsumoto, Nagano
  - Novartis Investigative Site, Nagano, Nagano
  - Novartis Investigative Site, Suwa, Nagano
  - Novartis Investigative Site, Ōmura, Nagasaki
  - Novartis Investigative Site, Nagaoka, Niigata
  - Novartis Investigative Site, Beppu, Oita Prefecture
  - Novartis Investigative Site, Uruma, Okinawa
  - Novartis Investigative Site, Habikino, Osaka
  - Novartis Investigative Site, Izumi, Osaka
  - Novartis Investigative Site, Moriguchi, Osaka
  - Novartis Investigative Site, Suita, Osaka
  - Novartis Investigative Site, Saga, Saga-ken
  - Novartis Investigative Site, Fukaya, Saitama
  - Novartis Investigative Site, Kawagoe, Saitama
  - Novartis Investigative Site, Tokorozawa, Saitama
  - Novartis Investigative Site, Hikone, Shiga
  - Novartis Investigative Site, Iwata, Shizuoka
  - Novartis Investigative Site, Shimotsuke, Tochigi
  - Novartis Investigative Site, Bunkyo Ku, Tokyo
  - Novartis Investigative Site, Higashimurayama, Tokyo
  - Novartis Investigative Site, Itabashi Ku, Tokyo
  - Novartis Investigative Site, Itabashi-ku, Tokyo
  - Novartis Investigative Site, Meguro City, Tokyo
  - Novartis Investigative Site, Minato-ku, Tokyo
  - Novartis Investigative Site, Nerima City, Tokyo
  - Novartis Investigative Site, Ōta-ku, Tokyo
  - Novartis Investigative Site, Shinagawa Ku, Tokyo
  - Novartis Investigative Site, Shinagawa-ku, Tokyo
  - Novartis Investigative Site, Shinjuku Ku, Tokyo
  - Novartis Investigative Site, Toyama, Toyama
  - Novartis Investigative Site, Tanabe, Wakayama
  - Novartis Investigative Site, Kofu, Yamanashi
  - Novartis Investigative Site, Fukushima
  - Novartis Investigative Site, Kagoshima
  - Novartis Investigative Site, Kumamoto
  - Novartis Investigative Site, Kyoto
  - Novartis Investigative Site, Niigata
  - Novartis Investigative Site, Osaka
  - Novartis Investigative Site, Shizuoka

IPD SHARING:
Plan to Share IPD: No